CLINICAL TRIAL: NCT03487224
Title: Neural Mechanisms of Decision Making in Hoarding Disorder
Acronym: LOSS
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Other Study IDs: 42327
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hoarding Disorder
Keywords: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hoarding Disorder: Adults diagnosed with Hoarding Disorder
  Interventions: Device: MRI with fMRI frequency
- Healthy Controls: Adults without mental illness
  Interventions: Device: MRI with fMRI frequency

INTERVENTIONS:
Device: MRI with fMRI frequency — Functional magnetic resonance imaging or fMRI measures brain activity by detecting changes in blood flow. Participants will do cognitive tasks during fMRI.

SUMMARY:
The purpose of this study is to understand the neural mechanisms of decision making in hoarding disorder.

DETAILED DESCRIPTION:
Hoarding disorder is a common and disabling disorder that represents a significant public health problem. This study aims to build on current research on decision making by examining these processes in hoarding disorder.

ELIGIBILITY:
Identify inclusion criteria.

Inclusion criteria for participants diagnosed with HD:

1. ages 18-70
2. primary diagnosis of hoarding disorder
3. sufficient severity of hoarding symptoms
4. stable on psychotropic medications for 1 month prior to study enrollment
5. capacity to provide informed consent
6. ability to tolerate clinical study procedures

Inclusion criteria for healthy control participants:

1. ages 18-70
2. capacity to provide informed consent

Identify exclusion criteria.

Exclusion criteria for participants with HD:

1. psychiatric or medical conditions that make participation unsafe
2. pregnant or nursing females
3. concurrent use of any medications that might increase the risk of participation (e.g. drug interactions)
4. presence of metallic device or dental braces

Exclusion criteria for healthy control participants:

1. any current or lifetime psychiatric diagnosis
2. current or past use of psychotropic medication
3. pregnant or nursing females
4. major medical or neurological problem
5. presence of metallic device or dental braces

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Hoarding Disorder and Healthy Participants
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-07-08 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
BOLD signal | up to 90 minutes
  BOLD signal derived from fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- See also: Stanford Medicine Faculty Page — http://med.stanford.edu/profiles/carolyn-rodriguez?tab=bio
- See also: Rodriguez Lab Website — http://med.stanford.edu/rodriguezlab/